CLINICAL TRIAL: NCT00510848
Title: Hamstrings Autograft Versus Tibialis Allograft for Reconstruction of Anterior Cruciate Ligament: Randomized Clinical Trial With 2 Year Follow-up
Brief Title: Hamstrings Autograft Versus Tibialis Allograft for Reconstruction of Anterior Cruciate Ligament
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/154
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2014-12

CONDITIONS: Rupture of the Anterior Cruciate Ligament With Instability of the Knee Joint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Reconstruction with an autograft tendon (hamstrings)
  Interventions: Procedure: autograft tendon
- 2 (Experimental): Reconstruction with an allograft tendon (tibialis posterior)
  Interventions: Procedure: allograft tendon

INTERVENTIONS:
Procedure: autograft tendon — Reconstruction with an autograft tendon (hamstrings)
  Arms: 1
Procedure: allograft tendon — Reconstruction with an allograft tendon (tibialis posterior)
  Arms: 2

SUMMARY:
Patients suffering from a rupture of the anterior cruciate ligament (ACL) with instability of the knee joint are treated with an operative ACL-reconstruction: one group of patients with a reconstruction with an autograft tendon (hamstrings), the other group with a reconstruction with an allograft tendon (tibialis posterior). The same surgical technique, the same fixation technique and the same rehabilitation protocol will be used in both groups. Follow-up will be done during 2 years.

ELIGIBILITY:
Inclusion Criteria:

* isolated rupture of the anterior cruciate ligament with instability of the knee joint
* meniscal tear possible to suture
* partial meniscectomies

Exclusion Criteria:

* chronic laxity (more than 9 months)
* associated collateral laxity (grade III)
* subtotal or total meniscectomy
* infection or inflammatory disease of the knee joint
* large cartilage lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
X-ray, CT-scan, KT1000 | 12 months

SECONDARY OUTCOMES:
X-rays, CT-scan, KT1000 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verdonk, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Robbrecht C, Claes S, Cromheecke M, Mahieu P, Kakavelakis K, Victor J, Bellemans J, Verdonk P. Reliability of a semi-automated 3D-CT measuring method for tunnel diameters after anterior cruciate ligament reconstruction: A comparison between soft-tissue single-bundle allograft vs. autograft. Knee. 2014 Oct;21(5):926-31. doi: 10.1016/j.knee.2014.05.003. Epub 2014 May 20. PMID 25022839